CLINICAL TRIAL: NCT03451734
Title: Optimizing and Individualizing the Pharmacological Treatment of First-episode Schizophrenic Patients
Status: Completed | Type: Observational
Sponsor: Central South University (Other)
Collaborators: Xiangya Hospital of Central South University (Other); Shanghai Mental Health Center (Other); West China Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); Air Force Military Medical University, China (Other); Jiangsu Province Nanjing Brain Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); Shanxi Medical University (Other); First Affiliated Hospital of Kunming Medical University (Other); Guangzhou Mental Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); Capital Medical University (Other); China Medical University, China (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Hebei Medical University (Other); Shenzhen Mental Health Center (Other); Sun Yat-sen University (Other); Wuhan Mental Health Centre (Other); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Renrong Wu,PhD, M.D,Ph.D,Professor, Central South University
Other Study IDs: 2016YFC1306900
Record Dates: First submitted 2018-01-23; First posted 2018-03-02 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Schizophrenia; Metabolic Syndrome
Keywords: Optimized and individualized antipsychotic treatment; Side Effect; Efficacy; Biomarker
MeSH Terms: conditions — Schizophrenia; Metabolic Syndrome | interventions — Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood,serum.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- treatment cohort: in sub-project 1, participants are randomized into olanzapine, risperidone, aripiprazole, amisulpride, ziprasidone, and haloperidol groups, we give them evaluation, and adjust dose of medication and deal with side effect if necessary.
  Interventions: Drug: antipsychotic medications
- adjunctive group: Patients who do not have an ideal response to antipsychotics treatment (reduction rate of Positive and Negative Symptom Scale (PANSS) score less than 25%) in sub-project 2 are recruited in this trial. They are randomly assigned to antipsychotic plus placebo, antipsychotic plus sulforaphane(3 tables per day, consisting of 30 mg of SFN-glucosinolate per day), and antipsychotic plus minocycline(200mg per day) groups, and the antipsychotic drugs used at this stage are still consistent with the first trial of sub-project 2. At baseline, 4 weeks and 8 weeks after treatment, all participants receive evaluations.
  Interventions: Drug: adjunctive group
- metformin and lifestyle intervention for MetS: Participants who develop MetS at the last visit in sub-project 1 and sub-project 2 are recruited in this trial. Patients are randomized into low-dose metformin (1000 mg/d), high-dose metformin (1500 mg/d), low dose metformin plus lifestyle intervention group (1000 mg/d), high dose metformin plus lifestyle intervention (1500 mg/d), lifestyle intervention, and placebo groups. The timepoints of the visits are at baseline, the 4th week, the 8th week, and the 12th week.
  Interventions: Drug: metformin and lifestyle intervention
- metformin and lifestyle prevention for high risk of MetS: Participants who are at a high risk of MetS are recruited in this trial. Participants are randomized into low dose metformin (750 mg/d), high dose metformin (1000 mg/d), lifestyle intervention, and placebo groups. The timepoints of the visits are at baseline, the 4th week, the 8th week, and the 12th week.
  Interventions: Drug: metformin and lifestyle intervention
- validation cohort: in sub-project 2, there are1,800 first-episode schizophrenia patients recruited from 19 hospitals, and six groups as with sub-project 1. The assessments (timepoint and content) are conducted as in sub-project 1.
  Interventions: Drug: antipsychotic medications

INTERVENTIONS:
Drug: antipsychotic medications — olanzapine, risperidone, aripiprazole, amisulpride, ziprasidone, and haloperidol groups
  Groups: treatment cohort; validation cohort
Drug: adjunctive group — antipsychotic plus placebo, antipsychotic plus sulforaphane(3 tables per day, consisting of 30 mg of SFN-glucosinolate per day), and antipsychotic plus minocycline(200mg per day) groups.
  Groups: adjunctive group
Drug: metformin and lifestyle intervention — different dose metformin combines lifestyle intervention
  Groups: metformin and lifestyle intervention for MetS; metformin and lifestyle prevention for high risk of MetS

SUMMARY:
The study is performed in 20 different hospitals from 19 cities in China. Three sub-projects are included. About sub-project 1, we build a clinical database system and a biological sample bank for data and samples management, which is applicable in other hospitals in this project. 1800 first-episode schizophrenia patients will be recruited in 19 sites and randomized into 6 treatment groups (olanzapine, risperidone, aripiprazole, ziprasidone, amisulpride, haloperidol). Through 8-week treatment and follow-up, we collect multidimensional indexes from psychopathology, neuropsychology, brain imaging, physiology, biochemistry, and life stress data. The summarized data is analyzed to screen potential biomarkers or biomarker panel that may predict the antipsychotic response, and ultimately to establish a prediction model.Sub-project 2, as an extension of sub-project 1, includes verification of the prediction model established in sub-project 1 and optimization of the current therapy with add-on treatment. Firstly, the validation process of the prediction model undergoes with an independent patient cohort. Next, we apply the add-on treatment to the patients who don't have ideal response to antipsychotic treatment after 8-week treatment. According to the results above, we manage to construct an optimized and individualized therapy for schizophrenia.In the end,We tend to conduct a randomized double-blind controlled trial to assess the safety and efficacy of the combination strategy for antipsychotic-induced metabolism syndrome, which includes metformin and lifestyle intervention. In the meanwhile, for schizophrenia patients at high-risk of metabolic syndrome, we tend to establish a prevention strategy expected to reduce or delay the occurrence of metabolic syndrome, which includes low-dose metformin and lifestyle intervention. We hope to successfully construct a comprehensive intervention strategy on metabolic syndrome induced by antipsychotic medications.

DETAILED DESCRIPTION:
For sub-project1 and 2:Inclusion criteria: Participants are ineligible to enter the trial under the following conditions: 1) Participants must be aged 18 to 65 years old who meet the criteria for schizophrenia diagnosed by Diagnostic and Statistical Manual of Mental Disorders-fifth edition (DSM-5) or International Classification of Diseases- tenth edition (ICD-10); 2) participants are in current episode of psychotic symptoms with a disease course less than 3 years and intermission less than 6 months; 3). there is at least 1 guardian to accompany patient within 1 year; 4). Participants and their guardians must sign an Informed Consent Form (ICF) indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion criteria (any potential paticipant who meets any of the following criteria will be excluded from participating in the study): 1). Participants with known or suspected clinically unstable systemic medical disorder; 2). participant has a current or prior DSM-5/ ICD-10 diagnosis of substance use disorder, intellectual disability, autism spectrum disorder, dementia or severe cognitive impairment; 3). planning to be pregnant, pregnancy or breast-feeding; 4). currently enrolled in another clinical trial.

For sub-project 3:The diagnostic criteria for Paticipants who develop metabolic syndrome: A. body mass index ≥ 25.0kg / m2; B. hyperglycemia: fasting blood glucose ≥ 110mg/dl (6.1mmol/l) and / or plasma glucose ≥ 140mg/dl(7.8mmol/l) after glucose load; and / or those who have been diagnosed with diabetes and received treatment; C. hypertension: systolic blood pressure (SBP) / diastolic blood pressure (DBP) ≥ 140/90mmHg, and / or those who have been diagnosed as hypertension and received treatment; D. dyslipidemia: at fasting state, total cholesterol (TG) ≥ 150 mg/dl (1.7mmol/l); and / or HDL-C: male < 35mg/dl (0.9mmol/l), female < 39mg/dl (1.0mmol/l) . The inclusive criteria for patients at high-risk of MetS: A. paticipants are taking antipsychotic drugs that significantly affect metabolisms, such as olanzapine, clozapine or risperidone; B. paticipants have family history of diabetes, hypertension and heart disease; C. the age of paticipants is over 40 years old; D. paticipants have no nonalcoholic fatty liver and gout; E. paticipants who have one or two components of metabolic syndrome but do not meet the diagnostic criteria.

For clinical and biological data collection, we collect blood samples and case information, which contains demographic data, medical history (including current medical history, past history, personal history and family history), medication regimen and results of follow-up evaluation. The biological samples are stored using unique code whose storage information can be linked to research case in the web server.

The Standard Operations Procedures (SOPs) are followed for data collection, storage, tracking, and utilization.

Professional technicians are employed for the establishment and subsequent maintenance of Internet platform, including web server and mobile terminal applications (APP). Ancillary researchers are involved for collection and timely upload of case information online. Principal investigators are responsible for auditing the data and quality control.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the Diagnostic and Statistical Manual (DSM-V) diagnostic criteria for schizophrenia;
2. Duration of illness less than 3 years with current symptoms exacerbation;
3. Male and female with aged 17 to 65 years;
4. Signed the study consent for participation

Exclusion Criteria:

1. Having history of substance dependence or abuse or whose symptoms are caused by the other diagnosable mental disorders;
2. Having history of traumatic brain injury, seizures or other known neurological or organic diseases of the central nervous system;
3. Taking antidepressants, stimulants, mood stabilizer or accepts electricity shock treatment;
4. Having current suicidal or homicidal thoughts or any safety concern by research staff that cannot be manage in an inpatient setting;
5. The routine blood tests showing abnormal renal, liver function;
6. Pregnant or lactating women.
7. No administration of any antibiotics in a mouth

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Meet the Diagnostic and Statistical Manual (DSM-V) diagnostic criteria for schizophrenia;Duration of illness less than 3 years with current symptoms exacerbation;Male and female with aged 17 to 65 years;
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Positive And Negative Syndrome Scale (PANSS) | 8 weeks
  The change of Positive And Negative Syndrome Scale (PANSS) total, positive and negative symptoms before and after treatment at different follow up point.
Clinical Global Impressions(CGI) | 8 weeks
  The change of Clinical Global Impressions(CGI):severity of illness(SI), global improvement(GI) and efficacy index(EI) before and after treatment at different follow up point.
Global Assessment Function(GAF) | 8 weeks
  The change of Global Assessment Function(GAF) before and after treatment at different follow up point.
MATRICS Consensus Cognitive Battery (MCCB) composite score | 8 weeks
  The investigators will use the MATRICS Consensus Cognitive Battery (MCCB) Composite score as primary cognitive outcome measure before and after treatment at different follow up point.

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Institute of 2nd Xiangya Hospital,CSU, Changsha, Hunan, China

REFERENCES:
- [Derived] Gao S, Xu Q, Han Y, Jiang J, Wu F, Peng T, Ling C, Ni S, Zhang R, Ming Y, Liu X, Xu X. Relationship between cognitive impairments and psychopathological symptoms in female schizophrenia subsequent to 8 weeks treatment with antipsychotic drugs. BMC Psychiatry. 2025 Mar 7;25(1):211. doi: 10.1186/s12888-025-06605-w. PMID 40055632
- [Derived] Xie P, Shao T, Long Y, Xie W, Liu Y, Yang Y, Huang Y, Wu R, Deng Q, Tang H. Orlistat for the treatment of antipsychotic-induced weight gain: an eight-week multicenter, randomized, placebo-controlled, double-blind trial. Lipids Health Dis. 2024 Jul 24;23(1):225. doi: 10.1186/s12944-024-02214-w. PMID 39049073
- [Derived] Zeng J, Zhang W, Lu X, Zhou H, Huang J, Xu Z, Liao H, Liang J, Liang M, Ye C, Sun T, Hu Y, She Q, Chen H, Guo Q, Yan L, Wu R, Li Z. The association of SOD and HsCRP with the efficacy of sulforaphane in schizophrenia patients with residual negative symptoms. Eur Arch Psychiatry Clin Neurosci. 2024 Aug;274(5):1083-1092. doi: 10.1007/s00406-023-01679-7. Epub 2023 Sep 20. PMID 37728803
- [Derived] Long Y, Wu Q, Yang Y, Cai J, Xiao J, Liu Z, Xu Y, Chen Y, Huang M, Zhang R, Xu X, Hu J, Liu Z, Liu F, Zheng Y, Meng H, Wang Z, Tang Y, Song X, Chen Y, Wang X, Liu T, Wu X, Fang M, Wan C, Zhao J, Wu R. Early non-response as a predictor of later non-response to antipsychotics in schizophrenia: a randomized trial. BMC Med. 2023 Jul 19;21(1):263. doi: 10.1186/s12916-023-02968-7. PMID 37468932
- [Derived] Xiao J, Huang J, Long Y, Wang X, Wang Y, Yang Y, Hei G, Sun M, Zhao J, Li L, Shao T, Wang W, Kang D, Liu C, Xie P, Huang Y, Wu R, Zhao J. Optimizing and Individualizing the Pharmacological Treatment of First-Episode Schizophrenic Patients: Study Protocol for a Multicenter Clinical Trial. Front Psychiatry. 2021 Feb 25;12:611070. doi: 10.3389/fpsyt.2021.611070. eCollection 2021. PMID 33716817
- [Derived] Peng XJ, Hei GR, Li RR, Yang Y, Liu CC, Xiao JM, Long YJ, Shao P, Huang J, Zhao JP, Wu RR. The Association Between Metabolic Disturbance and Cognitive Impairments in Early-Stage Schizophrenia. Front Hum Neurosci. 2021 Feb 22;14:599720. doi: 10.3389/fnhum.2020.599720. eCollection 2020. PMID 33692676
- [Derived] Huang J, Hei GR, Yang Y, Liu CC, Xiao JM, Long YJ, Peng XJ, Yang Y, Zhao JP, Wu RR. Increased Appetite Plays a Key Role in Olanzapine-Induced Weight Gain in First-Episode Schizophrenia Patients. Front Pharmacol. 2020 May 22;11:739. doi: 10.3389/fphar.2020.00739. eCollection 2020. PMID 32528286